CLINICAL TRIAL: NCT06576999
Title: Sensor-based Balance Training With Exergaming Feedback in Patients With Chronic Stroke
Brief Title: Sensor-based Balance Training With Exergaming Biofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE/PROG.60
Record Dates: First submitted 2024-08-20; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Stroke, Ischemic
Keywords: Chronic Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Randomised clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensor-based balance training (Experimental): The sensor-based balance training is performed using an integrated system composed of five inertial measurement units (IMUs) and a force platform. The system analyze the data via a notebook and provide a real-time feedback for the patient in a 32 inch screen in form of exergaming.
  Interventions: Device: Sensor-based Balance Training
- Usual balance training (Active Comparator): The usual balance training is performed using a series of conventional balance exercises administered by a formed physiotherapist that provided a verbal feedback about the quality of execution.
  Interventions: Other: Usual Balance Trainging

INTERVENTIONS:
Device: Sensor-based Balance Training — 10 sessions of sensor-based balance training with exergaming feedback. For this training an adaptive integrated audio-visual feedback system composed of five IMUs and a force platform connected wirelessly to a computer has been used. The training protocol include exercises of balance control, encompassing a total of five distinct exercises: i) Latero-lateral load shifting while seated; ii) Load shifting while standing: latero-lateral and antero-posterior, to simulate the balance control performed during the day; iii) Load control during sit-to-stand; iv) Gait swing and loading phase response: to stimulate a correct load shifting during the swing and stance phase; v) Latero-lateral load shifting with knee flexion.
  Other Names: SBT
  Arms: Sensor-based balance training
Other: Usual Balance Trainging — 10 sessions of usual balance training. The training includes: gait control exercises, weight shifting, and relies on both stable surfaces (i.e., steps) and unstable surfaces (i.e., oscillating platforms and various-sized fitballs). The protocol encompassed the application of stabilization techniques and the reaching of targets with the upper limb during upright position emulating the activity of daily living.
  Other Names: UBT
  Arms: Usual balance training

SUMMARY:
The purpose of this study is to evaluate the effects of a sensor-based balance training with exergaming feedback on balance skills in chronic stroke patients.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability globally, with many survivors experiencing persistent balance impairments that affect the quality of their life. In this context, the use of balance-focused rehabilitation might represent a promising strategy over traditional methods. The integration of biofeedback and advanced technology in rehabilitation, such as audiovisual feedback, can enhance cortical activation, sensory integration, and patient engagement. Exergaming, a specific form of biofeedback, exhibits potential in improving functional recovery and motivation in stroke rehabilitation. In fact, visual feedback has shown effectiveness in chronic stroke patients. Given the rising incidence of stroke and the associated challenges, it is crucial to explore new intervention strategies that leverage technological advancements for better balance recovery. Previous studies have shown promising results in subacute stroke patients using an integrated biofeedback system that combine inertial measurement units (IMUs) and a sensorized force platform. The current study aims to evaluate the effects of sensor-based training with exergaming feedback on balance functions in individuals with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Single event of cortical/subcortical ischemic stroke.
2. Onset > 180 days.
3. Lesion confirmed thought magnetic resonance (MR) or computer tomography (CT).
4. Able to stand upright with supervision or minimal assistance.

Exclusion Criteria:

1. Severe general impairment or concomitant diseases (i.e., Parkinson disease).
2. Orthopaedic contraindications.
3. Cognitive impairment (MINI MENTAL STATE EXAMINATION < 23).
4. Diagnosis of unilateral spatial neglect.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
The Berg Balance Scale (BBS) | Before training (t0); after 4 weeks of treatment (t1); after 8 weeks from the baseline (t2)
  The BBS is a clinical scale used to quantitatively assess balance ability after stroke. Range score from 0 to 56 points, a higher score represents an improvement.
The Canadian Neurological Scale (CNS) | Before training (t0); after 4 weeks of treatment (t1); after 8 weeks from the baseline (t2)
  The CNS is a clinical scale used to quantitatively assess neurological status of stroke patients. Range score from 1.5 to 11.5, a higher score represents an improvement.
The National Institutes of Health Stroke Scale (NIHSS) | Before training (t0); after 4 weeks of treatment (t1); after 8 weeks from the baseline (t2)
  The NIHSS Clinical scale used to quantitatively assess neurological status of stroke patients. Range score from 0 to 42, a lower score represents an improvement.
The Barthel Index (BI) | baseline (t0); 4weeks (t1 - end of treatment); 8weeks (t2 - 1 month follow-up)
  The BI is a clinical scale used to quantitatively assess functional independence after stroke. Range score from 0 to 100 points, a higher score represents an improvement.
The Rivermead Mobility Index (RMI) | Before training (t0); after 4 weeks of treatment (t1); after 8 weeks from the baseline (t2)
  The RMI is a questionnaire used to quantify mobility disability after stroke. Range score from 0 to 15 points, a higher score represents an improvement.
Postural stability | Before training (t0); after 4 weeks of treatment (t1); after 8 weeks from the baseline (t2)
  Postural stability has been recorded via a stabilometric platform to evaluate the oscillations of patients while standing in the upright position with open/closed eyes. The lenght of the Center of Pressure (CoP) has used to assess the change in postural stability. A reduction in the CoP represents an improvement.

OTHER OUTCOMES:
The Pittsburgh Rehabilitation Participation Scale (PRPS) | Recorded at the end of each session (10 sessions administered in 4 weeks)
  The PRPS is a clinician-rated instrument to assess participation of patients during therapies. Range score 1 to 6, a higher score represents higher motivation.

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Lucia Foundation, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
The datasets generated may be available from the corresponding author on reasonable request.